CLINICAL TRIAL: NCT00894725
Title: Laparoscopic vs. Open Left Colonic Resection: a Randomized Monocentric Trial
Brief Title: Laparoscopic Versus Open Left Colonic Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Marco Braga MD, San Raffaele Vita-Salute University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hmsxLPS09
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Colon Cancer; Benign Disease
Keywords: left colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LPS (Experimental): laparoscopic left colonic resection
  Interventions: Procedure: laparoscopic left colonic resection
- Open (Active Comparator): open left colonic resection
  Interventions: Procedure: open left colonic resection

INTERVENTIONS:
Procedure: laparoscopic left colonic resection — laparoscopic colonic resection
  Arms: LPS
Procedure: open left colonic resection — conventional open colonic resection
  Arms: Open

SUMMARY:
The main goal of this study is to clarify if laparoscopy (LPS) could become the standard approach in patients undergoing left colonic resection.

268 patient candidates to left colonic resection were randomly assigned to LPS (n=134) or open (n=134) approach. Postoperative care protocol was the same in both groups. Trained members of the surgical staff who were not involved in the study registered 30-day postoperative morbidity. Cost-benefit analysis was based on hospital costs. Long-term morbidity, quality of life, and 5-year survival have also been evaluated.

DETAILED DESCRIPTION:
The study design was explained to the potential participants who were asked to sign a written informed consent before randomization.

Eligible patients were randomly allocated to LPS or open surgery. Randomization list was computer generated. Assignments were made by means of sealed sequenced masked envelopes which were opened, before the induction of anesthesia, by a nurse unaware of the trial design.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* suitability to elective surgery

Exclusion Criteria:

* cancer infiltrating adjacent organs assessed by computed tomography
* cardiovascular dysfunction (New York Heart Association class > 3)
* respiratory dysfunction (arterial pO2 < 70 mmHg)
* hepatic dysfunction (Child-Pugh class C)
* ongoing infection
* plasma neutrophil level < 2.0x109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2000-02; Primary Completion 2004-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
short-term morbidity rate | 30 days

SECONDARY OUTCOMES:
long-term outcome | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, MD, Study Director — San Raffaele Vita-Salute University
Locations (1):
- San Raffaele Hospital, Surgical Department, Milan, Italy

REFERENCES:
- [Derived] Braga M, Frasson M, Zuliani W, Vignali A, Pecorelli N, Di Carlo V. Randomized clinical trial of laparoscopic versus open left colonic resection. Br J Surg. 2010 Aug;97(8):1180-6. doi: 10.1002/bjs.7094. PMID 20602506